CLINICAL TRIAL: NCT06827067
Title: Assessment of Effectiveness of Communication Skills and Anger Management Training Accompanied with Standardized Patient Given to Nurses
Brief Title: Communication Skills and Anger Management Training for Nurses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuksek Ihtisas University (Other)
Responsible Party: Principal Investigator, Arzu AYDOĞAN, Assistant Professor, Yuksek Ihtisas University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Dated 11/9/2016 and no. 15/10
Record Dates: First submitted 2025-01-29; First posted 2025-02-14 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Nurse-Patient Relations
Keywords: Difficult patient; Anger management; Communication; Simulation
MeSH Terms: conditions — Communication

STUDY DESIGN:
Intervention Model Description: A convergent parallel mixed-methods study design was used to address the questions comprehensively. In this study, randomized controlled trials were used quantitatively and a guided content analysis approach based on notes from debriefing sessions was used qualitatively. Quantitative data were evaluated with pre-test and post-tests.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (Other): Theoretical training consisting of a total of 7 sessions of 40-45 minutes each was given to 30 nurses in the control group.
  Interventions: Behavioral: Theoretical training
- Experimental group (Experimental): Immediately after the theoretical trainings of 30 nurses in the experimental group were completed, simulation trainings conducted with a standard patient were given. A half-day training was given to the standard patient (SH) about the scenario content before the application. Before the encounter with the SH, a preliminary interview was held with the nurses in the briefing room, where the content and purpose of the application were explained to the nurses, and the story of the SH was told to the nurses in line with the prepared scenario. Three nurses were interviewed for each scenario. The nurses communicated with the SH for 10-15 minutes and each interview was conducted using video recordings. Those who finished the interview with the SH watched the scenario of the other group as observers and at the end of each 3 scenarios, the debriefing phase lasting an average of 60-90 minutes was carried out.
  Interventions: Behavioral: Simulation application with standard patient; Behavioral: Theoretical training

INTERVENTIONS:
Behavioral: Simulation application with standard patient — Before the encounter with the standard patient (SH), a preliminary interview was held with the nurses in the briefing room, where the content and purpose of the application were explained to the nurses, and the story of the SH was told to the nurses in line with the prepared scenario. Three nurses were interviewed for each scenario. The nurses communicated with the SH for 10-15 minutes and each interview was conducted using video recordings. Those who finished the interview with the SH watched the scenario of the other group as observers, and at the end of each 3 scenarios, the debriefing phase was carried out for an average of 60-90 minutes.
  Arms: Experimental group
Behavioral: Theoretical training — The trainings, each of which lasted 40-45 minutes on average, were conducted in a total of 7 sessions.

SUMMARY:
Objective: The aim of this study was to determine the effect of training given to nurses on communication and anger management skills in the presence of standardized patients.

Method: The study was conducted using a convergent parallel design, which is a mixed-method design. The experimental and control groups of the study were conducted with a total of 56 nurses. Data were collected using a socio-demographic data collection form, Communication Skills Inventory and State-Trait Anger and Anger Expression Scale. The intervention group participated in the simulation, and qualitative data were collected during the debriefing session of the simulation. The scales were administered to the groups 3 times in total: before the training, after the training and 6 weeks after the end of the training.

DETAILED DESCRIPTION:
The patient-nurse relationship is a dynamic process that can change as the patient's health needs change and nurses can show positive emotions and behaviors to their patients. However, due to the nature of human beings, it may be impossible to show positive behaviors at all times, and in communication processes, situations that make communication difficult may occur from time to time (Gorman 1996). When the studies examining the communication between patients and nurses are examined, it is found that some patient behaviors that may cause problems in the relationship and the inadequacies of nurses in controlling their emotions are the causes. When these studies are examined, the concept of "difficult patient" attracts the most attention (Akgün-Çıtak 2011, Wolf and Smith 2007, Macdonald 2007, Kennedy Sheldon et al. 2006).

"Difficult patients" are defined in the literature as patients with behaviors that hinder communication. (Göral 2011, Koekkoek et al. 2006). In a study conducted by Essary et al. (2005), it was observed that patients were labeled as "difficult patients" as a result of ineffective communication between nurse and patient and that nurses tended to blame patients as a result of labeling. In the literature, it is stated that improving communication skills with the difficult patient group will benefit nurses and the onset of conflicts can be prevented, which should not be forgotten that conflicts that cannot be prevented arouse feelings of anger in individuals. (MacLean at all 2017, Baran and Okanlı 2015) For this reason, it is as important for nurses to improve their communication skills as it is for them to improve their ability to cope with anger.

Although anger is a frequently felt emotion in the nursing profession, this emotion should not be expressed with aggression or suppressed in order to be healthy and useful. Nurses should gain the ability to express anger in a healthy way by recognizing and accepting it like all other emotions (Bozkurt 2010, Akdeniz 2007). Expressing anger openly in an acceptable way is a positive personality trait. However, such emotions that cannot be controlled and are ignored by denial or suppression have the potential to be harmful for both the person and his/her environment (Kaya et al. 2012). In the study conducted by Baran and Okanlı in 2015, it was emphasized that nurses should regularly receive in-service trainings on anger and anger expression in order to recognize their anger, accept its existence and express their anger correctly. Trainings on anger management can be given in many ways like other trainings. These ways can be in the form of individual and group trainings as well as using various simulations.

Simulation-based trainings are ideal for nursing education as they include an interactive method that can be used to teach cognitive, psychomotor or emotional skills to individuals or groups at any skill or proficiency level. ( Zengin & Eren Fidancı 2024, Tanis, Quinn, & Bischoff, 2019) In standardized patient simulation, the patient or case study is animated by playing the scenario prepared with structured steps. The use of standardized patients in teaching contributes to the development of participants' communication skills, history taking and physical examination skills. ( Zengin & Eren Fidancı 2024). When the literature is examined, it is seen that skill-oriented studies are frequently used in simulation-based studies, but emotion-oriented studies are weaker, and the majority of the studies are conducted with student nurses, and the intervention study conducted with working nurses is very limited.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the research
* Working as a nurse in any of the surgical or internal medicine clinics of the hospital
* According to the results of the pre-test application, anger control scores were lower than the other nurses participating in the study.

Exclusion Criteria:

* Not volunteering to participate in the study
* Not having participated in simulation training in the experimental group

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2018-02-13 (Actual)

PRIMARY OUTCOMES:
State-Trait Anger and Anger Expression Scale | Measurements taken just before the training begins.
  State-Trait Anger and Anger Expression Scale is a self-assessment scale that measures the feeling and expression of anger. The State-Trait Anger and Anger Expression Scale , developed by Spielberger (1983) and whose Turkish validity and reliability were determined by Özer (1994), consists of 4 sub-dimensions and 34 items, namely anger-in, anger-out, anger control, and trait anger. Participants were asked to respond using a 4-point Likert-type scale (1 "Does not describe at all," 2 "Somewhat describe," 3 "Fairly describe," and 4 "Completely describe"). High scores on the trait anger dimension indicate that the level of anger is high, high scores on the anger control dimension indicate that anger can be controlled, high scores on the anger-out dimension indicate that anger is easily expressed, and high scores on the anger-in dimension indicate that anger is suppressed.
Communication Skills Inventory | Measurements taken just before the training begins.
  Inventory developed by Balcı and Ersanlı (1998) to measure the level of communication skills among university students. The scale consists of three sub-dimensions including behavioral, cognitive and emotional. The scale consists of a total of 10 items. There are 15 items that measure each dimension. The scale has been developed in the 5-point Likert type. The highest score that can be achieved from the scale is 225, and the lowest score is 45. Correlation between the total score from Communication Skills Inventory and total scores of each dimension was found to be 0.85 for intellectual sub-dimension, as 0.73 for emotional sub-dimension and 0.82 for behavior sub-dimension. Regarding the validity study of the inventory; its correlation with Communication Skills Assessment Scale developed by Korkut (1996) was examined. In the validity study carried out, correlation coefficient between two scales was found as 0.70. This value is thought to be enough for the validity of the scale.

SECONDARY OUTCOMES:
State-Trait Anger and Anger Expression Scale | Immediately after the trainings
  After the theoretical trainings were completed, State-Trait Anger and Anger Expression Scale forms were applied to the control group and their scores were evaluated after the training. The scales were applied to the experimental group immediately after the simulation training was completed and their scores were evaluated.
Communication Skills Inventory | Immediately after the trainings
  After the theoretical trainings were completed, Communication Skills Inventory forms were applied to the control group and their scores were evaluated after the training. The scales were applied to the experimental group immediately after the simulation training was completed and their scores were evaluated.

OTHER OUTCOMES:
State-Trait Anger and Anger Expression Scale | Six weeks after the trainings are completed
  Six weeks after the completion of all trainings, the experimental and control groups were administered the State-Trait Anger and Anger Expression Scale for the third time.
Communication Skills Inventory | Six weeks after the trainings are completed
  Six weeks after the completion of all trainings, the experimental and control groups were administered the Communication Skills Inventory for the third time.

CONTACTS AND LOCATIONS:
Overall Officials: Arzu AYDOĞAN, Principal Investigator — Yuksek Ihtisas University
Locations (1):
- Yuksek Ihtisas University, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Study data may be shared upon request within the scope of data privacy